CLINICAL TRIAL: NCT05915572
Title: Effect of Mulligan Technique on Shoulder Dysfunction Post Neck Dissection Surgeries
Brief Title: Mulligan Technique on Shoulder Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Amin Ziethar, Assistant Lecturer at Department of Surgery and Burn - Faculty of Physical Therapy - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 752015
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Cancer
Keywords: Mulligan Technique; Shoulder Dysfunction; Neck Dissection Surgeries
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization Technique Plus Traditional Physical Therapy Program (Experimental): Mulligan Mobilization Technique plus traditional physical therapy program 3 sessions per week for 6 weeks.
  Interventions: Other: Mulligan Mobilization Technique; Other: Traditional Physical Therapy Program
- Traditional Physical Therapy Program (Experimental): Traditional physical therapy program 3 sessions per week for 6 weeks
  Interventions: Other: Traditional Physical Therapy Program

INTERVENTIONS:
Other: Mulligan Mobilization Technique — The therapist applied passive accessory glide to increase shoulder flexion, abduction, external rotation
  Arms: Mulligan Mobilization Technique Plus Traditional Physical Therapy Program
Other: Traditional Physical Therapy Program — Myofascial release and ROM ex. 3 sessions per week for 6 weeks.

SUMMARY:
76 patients suffering from shoulder dysfunction following neck dissection surgeries will participate in this study. The participants will be selected from Damanhur Oncology Center and randomly will be distributed into two groups.

Group (A): 38 patients will receive MWM in plus traditional physiotherapy program 3 sessions per week for 6 weeks.

Group (B): 38 patients will receive traditional physiotherapy program 3 sessions per week for 6 weeks.

DETAILED DESCRIPTION:
1) Subjects: 76 patients suffering from shoulder dysfunction following neck dissection surgeries will participate in this study. The participants will be selected from Damanhur Oncology Center and randomly will be distributed into two groups.

Group (A): 38 patients will receive MWM in plus traditional physiotherapy program 3 sessions per week for 6 weeks.

Group (B): 38 patients will receive traditional physiotherapy program 3 sessions per week for 6 weeks.

The participants will be selected from Damanhur Oncology Center and randomly will be distributed into two groups equal in number.

2) Equipment:

Therapeutic equipment:

* Mulligan Mobilization Technique: to increase shoulder flexion, abduction, external rotation
* Traditional physical therapy program:

Measurement equipment:

* Digital Goniometer
* Shoulder Pain and Disability Index

ELIGIBILITY:
Inclusion Criteria:

* Patients' age will be between 30-50 years old.
* Both gender 76 patients will participate in this study.

Exclusion Criteria:

* Patients with rotator cuff tears and other shoulder ligament injuries or tendon calcification.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Digital Goniometer | 6 weeks
  Measure shoulder ROM

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index | 6 weeks
  Measure pain and disability

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethical Committee Faculty of Physical Therapy, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt